CLINICAL TRIAL: NCT05476835
Title: Effect of Pulmonary Rehabilitation Program on Post Hospitalization Severe COVID- 19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Enas Sayed Farhat, Fayoum University Hospital, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no: 170 session 82
Record Dates: First submitted 2022-07-23; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Intervention Model Description: 50 patients were enrolled in the study post hospitalization due to severe COVID 19 infection. Dyspnea score, Spirometry and 6minute walk test were performed upon discharge. Pulmonary rehabilitation program was performed. Follow up assessment of the same parameters was done 6 weeks after the program.
  These results were compared with another 50 patients who were admitted in hospital due to severe COVID 19 infection but no pulmonary rehabilitation program was performed to them after hospitalization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (group A) - control group (groupB) (Experimental): The experimental group (group A) performed respiratory exercises (in form of diaphragmatic breathing, pursed lip breathing exercise and incentive spirometer), rehab exercise program and walking exercise.
  Interventions: Combination Product: respiratory exercises - incentive spirometer - walking
- control group (group B) (No Intervention): The control group (group B) did not receive any physical therapy program

INTERVENTIONS:
Combination Product: respiratory exercises - incentive spirometer - walking — respiratory exercises (in form of diaphragmatic breathing, pursed lip breathing exercise and incentive spirometer), rehab exercise program and walking exercise.
  Arms: experimental group (group A) - control group (groupB)

SUMMARY:
COVID-19 infection was discovered to be the major global cause of a serious respiratory illness toward the end of 2019. The majority of COVID-19 patients experience mild disease, while about 14% go on to have severe disease and 6% end up in critical condition. An evidence-based standard of therapy called pulmonary rehabilitation includes exercise training, education, and behavior modification to help people with lung illness feel better physically and mentally.

The aim of the study to evaluate the effect of pulmonary rehabilitation program on severe post covid19 patients (post hospitalization) regarding pulmonary function tests and dyspnea score.

DETAILED DESCRIPTION:
SARS CoV-2 infection has caused substantial death, morbidity, and unprecedented strain on the world's healthcare systems . When the illness is minor, it typically takes two weeks from the onset of symptoms till recovery, and when it is severe or critical, it may take three to six weeks. It should be mentioned that approximately 75% to 80% of hospitalized patients will remain there for more than 21 days .

After the virus is defeated, COVID-19 can have serious aftereffects on the patient, with bilateral pneumonia. As a result, physiotherapy is essential in this pandemic and will play a major role in helping many patients' health. A 20-30% reduction in pulmonary capacity has already been reported in recent studies .

Although pulmonary rehabilitation has been suggested following severe COVID-19, there is a lack of data showing effectiveness on recovery of physical and psychosocial parameters in severe COVID-19 patients following hospitalization.

The aim of the study is to evaluate the effect of pulmonary rehabilitation program on severe post covid19 patients (post hospitalization) regarding pulmonary function tests and dyspnea score.

50 patients were enrolled in the study post hospitalization due to severe COVID 19 infection. Dyspnea score, Spirometry and 6minute walk test were performed upon discharge. Pulmonary rehabilitation program was performed. Follow up assessment of the same parameters was done 6 weeks after the program.

These results were compared with another 50 patients who were admitted in hospital due to severe COVID 19 infection but no pulmonary rehabilitation program was performed to them after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 50 and 70 years.
* Severe COVID infection.
* Impaired pulmonary function tests post COVID infection.

Exclusion Criteria:

* Mild or moderate COVID infection.
* Normal pulmonary function tests post COVID infection
* Chronic chest disease
* End organ failure (sever heart disease-neurodegenerative disease- sever stroke)
* Unstable angina, myocardial infarction, angioplasty, heart surgery in the previous 3 months
* Chronic renal impairments.
* Epistaxis, active haemoptysis
* Recent facial, oral, or skull surgery or trauma.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
improvement in dyspnea scale | 6 weeks
  modified medical research council scale (mMRC)
improvement in spirometry measures | 6 weeks
  forced vital capacity measurement in spirometry

SECONDARY OUTCOMES:
improvement in oxygen saturation and 6 minute walk test | 6 weeks
  oxygen saturation before and after 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa M Younis, doctorate, Study Chair — Fayoum University Hospital
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
demographic data of patients - dyspnea scale - pulmonary function tests - oxygen saturation before and after study